CLINICAL TRIAL: NCT03080857
Title: Computer Simulated Atrial Fibrillation Tool to Reduce Hospitalizations and Emergency Department Visits
Brief Title: Computer Simulated Atrial Fibrillation Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Cardiac Arrhythmia Network of Canada (Other)
Responsible Party: Principal Investigator, Ratika Parkash, Staff Cardiologist, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RP-003
Record Dates: First submitted 2017-03-09; First posted 2017-03-15 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Cohort study to assess a computer simulated electronic platform
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Platform (Experimental): Patients will be provided with a computer simulated tool to assist with education and support relating to atrial fibrillation.
  Interventions: Other: Virtual Platform; Device: AliveCor Heart Monitor

INTERVENTIONS:
Other: Virtual Platform — The platform will direct patients to review the Canadian Cardiovascular Guidelines and the Heart & Stroke website for commonly asked questions relating to atrial fibrillation, as well as recommendations regarding nutrition and activity.
  Other Names: Computer simulated atrial fibrillation tool (CSAF Tool)
Device: AliveCor Heart Monitor — A substudy of patients enrolled into the CSAF Tool study who own a compatible smart phone will be randomized to the Alive Cor Heart Monitor plus the virtual platform versus the virtual platform alone. The purpose of this substudy is to assess the feasibility and effect of incorporating Alive COR into a virtual online patient-education platform on patients' quality of life and AF-related emergency room visits and hospitalizations.

SUMMARY:
This will be a before-after study, using a prospective cohort to evaluate the use of a virtual, patient-centered platform as compared to a historical cohort of patients with atrial fibrillation (AF) and if the education and support provided by the platform will reduce Emergency Department visits for AF.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common sustained arrhythmia affecting 1-2% of the population of the western world, increasing to 10% in patients above the age of 75. The lifetime risk for development of AF is 26% for men and 23% for women. It is associated with significant morbidity, mortality and cost, but also with a two-fold increase in mortality and a six-fold risk of stroke. Severity of symptoms for AF may range from a 'nuisance' feeling of palpitations to debilitating symptoms that affect quality of life, interfere with normal livelihood and significantly impair exercise tolerance to more severe symptoms (hemodynamic compromise and heart failure), which are associated with poor prognosis and increased mortality. Patients who are symptomatic pose the greatest burden to the health care system, often making repeated visits to the emergency room for treatment or repeated hospitalizations.

AF is known to be a chronic disease. The majority of patients have progressively more episodes of AF, or present with persistent AF. As with all chronic diseases, it cannot be cured but can be controlled with effective treatments. AF often occurs in the setting of other diseases, increasing the complexity in determining appropriate therapies. Most often, AF occurs in the setting of other cardiovascular disease, obesity, diabetes, sleep apnea or a combination of the above. In order to effectively manage AF, a 'holistic' approach is necessary. Appropriate management of hypertension, sleep apnea, obesity, etc. is part of the mainstay of therapy for AF. This is part of the Canadian Cardiovascular Society (CCS) AF guidelines recommendations stating: "underlying causes or precipitating factors for AF including hypertension should be identified and treated". Current guidelines suggest that AF treatment should focus on strategies to manage and control heart rate and rhythm. Exercise and physical activity have been shown to improve outcomes in patients with some cardiac conditions (ischemic heart disease, myocardial infarction, congestive heart failure), but its effects on AF are still not clear.

The current Canadian health care system was designed to address acute illness, rather than chronic disease, which is impacting hospitalizations for symptomatic AF. There is not an AF clinic at the QEII Health Sciences Centre to assist with AF management after a patient has been seen by a specialist. The investigators propose to create, evaluate, refine and implement a virtual, patient-centered platform to guide patients with out-of-hospital management of atrial fibrillation, after evaluation by a specialist.

ELIGIBILITY:
Inclusion Criteria:

* can ambulate independently
* provide informed consent
* have documented symptomatic AF
* are proficient in the English language
* have access to a computer, tablet or smartphone

Exclusion Criteria:

* unable to participate due to physical limitations
* are planning to move during the period of study
* have a medical condition making 1 year survival unlikely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of using the simulated AF clinic platform | 6 months
  Assessing the percentage of patients who utilize the virtual patient platform on a regular basis to guide their management. A successful pilot will be defined as: 90% of patients use the platform at least once, 75% of patients use it at least twice over the six month follow up period.

SECONDARY OUTCOMES:
Patient satisfaction | 6 months
  Semi-quantitative data will be collected regarding patient satisfaction with the platform.

CONTACTS AND LOCATIONS:
Overall Officials: Ratika Parkash, MD FRCPC, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- QE II Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No